CLINICAL TRIAL: NCT06678893
Title: Pilor Trial of Auricular Acupuncture for Latent Labor-Related Pain and Anxiety
Brief Title: Ear Acupuncture for Pain and Anxiety Management in Early Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Kalin Gregory-Davis, MD, Resident Physician, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2145161-3
Record Dates: First submitted 2024-10-29; First posted 2024-11-07 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Pain; Anxiety; Labor
Keywords: Acupuncture; Auricular Acupuncture; Early labor; Pain; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders; Obstetric Labor, Premature

STUDY DESIGN:
Intervention Model Description: This is a pilot study of a randomized control trial. Consented participants will be randomized to either auricular acupuncture or placebo intervention. Blood pressure, heart rate, and VAS pain and anxiety scores will be recorded and compared pre and post intervention in both treatment arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Auricular Acupunture (Experimental): Participants randomized to this arm will undergo treatment with the 5 Needle Protocol of Auricular Acupuncture
  Interventions: Device: Acupuncture Needle on an adhesive
- Placebo (Placebo Comparator): Participants randomized to this arm will undergo treatment with small adhesives without needles placed in the same configuration as the 5 Needle Protocol
  Interventions: Device: Adhesives

INTERVENTIONS:
Device: Acupuncture Needle on an adhesive — This study utilizes acupuncture needs on small adhesives which will be placed according to the 5NP NADA Auricular Acupuncture Protocol.
  Arms: Auricular Acupunture
Device: Adhesives — For those randomized to the placebo arm, adhesives without needles will be placed according to the 5NP NADA Auricular Acupuncture Protocol placement
  Arms: Placebo

SUMMARY:
This is a study evaluating the feasibility and acceptability of ear acupuncture for the management of pain and anxiety in early labor.

DETAILED DESCRIPTION:
This double blinded randomized controlled pilot study will take place in the Emergency Department of Women and Infants Hospital (WIH) in Providence Rhode Island. This study seeks to assess feasibility and acceptability utilizing the 5 Needle Protocol of Auricular Acupuncture (5NP, AA) during early labor for management of pain and anxiety. At the time of emergency department evaluation at Women and Infants Hospital for a chief complaint of painful contractions, the investigators will enroll 40 pregnant people as a feasibility sample investigating the impact of auricular acupuncture (AA) on patient-reported pain and anxiety in early labor. Participants will be randomized to either AA using the 5 Needle protocol versus placebo acupuncture. While the data on the efficacy of auricular acupuncture for pain and anxiety is mounting, evidence for utility in treating labor pain is limited. This proposal will be one of the first to randomize pregnant people presenting with concern for pain or anxiety related to labor contractions to this potential treatment.

The investigator's long-term goal is to find an effective treatment option for a common labor complaint while improving satisfaction with pain management in the Emergency Department. Given this is a pilot study, the primary objective is to determine feasibility of implementing a randomized control trial evaluating the effect of auricular acupuncture as an initial treatment for improving perceived pain and anxiety symptoms related to contractions. The central hypothesis is that this is indeed feasible and acceptable in the Emergency Department setting of Women and Infants Hospital in Rhode Island. The secondary objective is to assess the trend that auricular acupuncture has on pain and anxiety scores, as well as on heart rate and blood pressure. Though the sample size is aimed to assess feasibility and will not be sufficiently powered for an efficacy analysis, if trends suggest that auricular acupuncture decreases pain and/or anxiety sores, further investigation with a larger randomized control trial will be warranted.

Eligible participants for this trial include Spanish or English speaking patients 18 years or older who are in early labor with a singleton pregnancy greater than or equal to 37+0 weeks gestation, and willing to be randomized to receive auricular acupuncture versus placebo. Early labor will be defined as less than 6 centimeters dilated and experiencing at least 2 contractions in ten minutes, per patient report and/or tocometry. Exclusion criteria include patients less than 18 years of age, non-Spanish or English-speaking patients, multi-gestation, preterm labor, greater than or equal to 6 cm dilated, less than 2 contractions in 10 minutes, morphine or nitrous oxide administration within the last two hours, congenital anomalies, open wounds or skin disorders of the ear, previous adverse reactions to acupuncture and/or allergies or contraindications to adhesives.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, Spanish or English speaking, with term (37+ weeks pregnant) singleton pregnancy, in early labor (as defined as less than 6cm dilated and having at least 2 contractions in 10 minutes)

Exclusion Criteria:

* Younger than 18 years old, non-english or spanish speaking, greater than 6cm or not having consistent contractions (less than 2 contractions in 10 minutes), preterm and/or multiple gestation pregnancy, received morphine or nitrous oxide within the last 2 hours, congenital anomalies/wound/skin disorders of the ear, or prior adverse reaction to acupuncture, adverse reactions or allergies to adhesives.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Percent of eligible participants that consent to being a part of the study | up to 3 months
  The investigators are evaluating if doing a randomized control trial on acupuncture in early labor is feasible in the setting of the Emergency Department of Women and Infants Hospital in Rhode Island by evaluating how many eligible patients consent to being a part of the study
Likert scale 1 to 5 of patient satisfaction with treatment experience | up to 3 months
  We are evaluating if doing acupuncture during labor is acceptable to patients in the emergency department of Women and Infants Hospital by using a Likert scale questionnaire evaluating their experience of receiving the intervention and their likelihood of doing the intervention were it to be offered again. The lowest value of the scale is 1 and the highest is 5. A higher number indicates higher level of satisfaction with the intervention performed.

SECONDARY OUTCOMES:
Visual Analogue Scale pain score | 30 minutes
  The investigators are comparing visual analogue scale pain scores pre and post acupuncture versus placebo intervention to see if there is a reduction in pain score that correlates with our intervention. This study is not powered to prove causality but we will look for correlation as a secondary outcome. The minimum value on the scale is 0 and the maximum is 10. A higher number indicates higher levels of pain.
Visual Analogue Scale Anxiety Scores | 30 min
  The investigators will be evaluating visual analogue scale Anxiety scores pre and post intervention of placebo versus acupuncture to see if there is a reduction in anxiety that correlates with our intervention. This study is not powered to prove causality however will look for correlation as a secondary outcome. The minimum value on the scale is 0 and the maximum is 10. A higher number indicates higher levels of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Women and Infants Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
As of now, this is a single site feasibility study. If we move forward with a larger multi-center study, we will plan to share IPD but at this time, given it is a single site and feasibility study we do not have a plan to share IPD with anyone other than the key study personnel.

REFERENCES:
- [Background] Levett KM, Smith CA, Dahlen HG, Bensoussan A. Acupuncture and acupressure for pain management in labour and birth: a critical narrative review of current systematic review evidence. Complement Ther Med. 2014 Jun;22(3):523-40. doi: 10.1016/j.ctim.2014.03.011. Epub 2014 Apr 13. PMID 24906592
- [Background] Baumler P, Zhang W, Stubinger T, Irnich D. Acupuncture-related adverse events: systematic review and meta-analyses of prospective clinical studies. BMJ Open. 2021 Sep 6;11(9):e045961. doi: 10.1136/bmjopen-2020-045961. PMID 34489268
- [Background] Zhang CS, Yang AW, Zhang AL, May BH, Xue CC. Sham control methods used in ear-acupuncture/ear-acupressure randomized controlled trials: a systematic review. J Altern Complement Med. 2014 Mar;20(3):147-61. doi: 10.1089/acm.2013.0238. Epub 2013 Oct 19. PMID 24138333
- [Background] Vakilian K, Ghaemmaghami M, Sheikhganbari N, Shabani F, Vahedi M. Reducing Labor Anxiety with Auriculotherapy: A Randomized Clinical Trial Study. Chin J Integr Med. 2022 May;28(5):440-444. doi: 10.1007/s11655-021-3452-0. Epub 2021 Sep 28. PMID 34581941
- [Background] Smith CA, Collins CT, Levett KM, Armour M, Dahlen HG, Tan AL, Mesgarpour B. Acupuncture or acupressure for pain management during labour. Cochrane Database Syst Rev. 2020 Feb 7;2(2):CD009232. doi: 10.1002/14651858.CD009232.pub2. PMID 32032444
- [Background] King HC, Hickey AH, Connelly C. Auricular acupuncture: a brief introduction for military providers. Mil Med. 2013 Aug;178(8):867-74. doi: 10.7205/MILMED-D-13-00075. PMID 23929047
- [Background] Thomson G, Feeley C, Moran VH, Downe S, Oladapo OT. Women's experiences of pharmacological and non-pharmacological pain relief methods for labour and childbirth: a qualitative systematic review. Reprod Health. 2019 May 30;16(1):71. doi: 10.1186/s12978-019-0735-4. PMID 31146759
- See also: This is the website for the People's Organization of Community Acupuncture, this is the organization through which the key study personnel were trained in auricular acupuncture — https://pocacoop.com/
- See also: Providence Community Acupuncture is the local organization that hosted the training and education for our key study personnel to learn auricular acupuncture — https://pca-pins.com/